CLINICAL TRIAL: NCT02691936
Title: A Randomized Clinical Trial Comparing Vaginal Laser Therapy to Vaginal Estrogen Therapy in Women With Genitourinary Syndrome of Menopause
Brief Title: Comparison of Vaginal Laser Therapy to Vaginal Estrogen Therapy
Acronym: VeLVET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: Foundation for Female Health Awareness (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15-1570
Record Dates: First submitted 2016-02-22; First posted 2016-02-25 (Estimated); Results first posted 2019-10-17 (Actual); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: Atrophic Vaginitis; Menopause
Keywords: Genitourinary symptoms of menopause; Menopause; Atrophic vaginitis
MeSH Terms: conditions — Atrophic Vaginitis | interventions — Estrogens, Conjugated (USP)

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CO2 fractionated vaginal laser (Experimental): Postmenopausal women will undergo treatment intravaginally with the fractional microablative CO2 laser system MonaLisa Touch vaginal laser protocol x 3 time points at baseline, 6 weeks and 3 months.
  Interventions: Device: CO2 fractionated vaginal laser
- Estrogens, Conjugated (USP) (Active Comparator): The women in the vaginal estrogen group will be prescribed and asked to administer the conjugated estrogen cream 0.5 g of cream equivalent to 0.625 mg of conjugated estrogen.
  Interventions: Drug: Estrogens, Conjugated (USP)

INTERVENTIONS:
Device: CO2 fractionated vaginal laser — Intravaginal treatment with fractional microablative CO2 laser at baseline, 6 weeks and 3 months
  Other Names: MonaLisa Touch
  Arms: CO2 fractionated vaginal laser
Drug: Estrogens, Conjugated (USP) — Conjugated estrogen cream 0.5g (equivalent of 0.625 mg of conjugated estrogen) daily for two weeks then twice weekly for 24 weeks
  Other Names: Vaginal Estrogen cream
  Arms: Estrogens, Conjugated (USP)

SUMMARY:
This is a multi-centered, randomized prospective single blinded clinical trial comparing CO2 fractionated vaginal laser therapy and vaginal estrogen cream therapy in the treatment of vulvovaginal atrophy/GSM.

DETAILED DESCRIPTION:
This is a multi-centered, randomized prospective single blinded clinical trial comparing CO2 fractionated vaginal laser therapy and vaginal estrogen cream therapy in the treatment of vulvovaginal atrophy/GSM.

Subject Recruitment and Screening Study subjects will be recruited from patients who present to the clinical sites at the Women's Health Institute at the Cleveland Clinic, Christ Hospital, Stanford University Hospital, MedStar Washington Hospital Center, Women's and Infants' Hospital of Rhode Island and Wake Forest Baptist Medical Center for treatment of GSM. Cleveland Clinic will serve as the central Data Coordinating Center

Study Identification and Recruitment Potential subjects will be identified by members of the sections of Urogynecology and Reconstructive Pelvic Surgery and Benign Gynecology at the respective institutions. Eligible patients who agree to participate will be provided written informed consent administered by the collaborators listed on this IRB.

Randomization The participants will then be randomized to either fractional CO2 vaginal laser therapy or vaginal estrogen cream according to a computer-generated randomization schedule with random block sizes with the use of the SAS statistical software package (SAS Institute, Cary, NC). All patients will be unblinded to their assignment.

Diagnostic and Therapeutic Interventions In addition to a standardized evaluation including the history and physical examination, patients will be asked to complete the Female Sexual Function Inventory (FSFI) questionnaire, the Day-to-day Impact of Vaginal Aging (DIVA) questionnaire, and the Urogenital Distress Inventory (UDI-6), at baseline, 3 months, and 6 months after baseline and visual analog scales (VAS) for GSM symptoms. The Patient Global Index (PGI) will also be administered at 6 months. Completion of these questionnaires should take no more than 15-20 minutes. A vaginal maturation index will be obtained at the baseline visit on a regular Pap Smear side and fixed with cytofixative and air dried. This will be repeated during the last follow up visit at 6 months.

Vaginal Laser Protocol Postmenopausal women will undergo treatment intravaginally with the fractional microablative CO 2 laser system (SmartXide 2 V 2 LR, MonaLisa Touch, DEKA, Florence, Italy), using the following setting: dot power 30 watt, dwell time 1000 μ s, dot spacing 1000 μ m and the smart stack parameter from 1 to 3. Stack 1 is used at baseline and stack 3 at 6 weeks and 3 months. The laser beam will be applied using a 90° vaginal probe gently inserted up to the top of the vaginal canal and subsequently withdrawn at centimeter intervals and rotated to 6 positions in an alternating clockwise and counterclockwise pattern in order to provide a complete treatment of the vaginal wall. At the investigators discretion a flat probe (vulvar probe) may be utilized to more efficiently treat the introital area and vestibule. At the level of the vaginal introitus, the dot power will be decreased to 26 watts. A treatment cycle includes three laser applications (every 40-50 days, approximately 6 weeks). The procedure will be performed in the outpatient clinic and does not require any specific preparation (e.g. analgesia/anesthesia). At the clinician's discretion, EMLA cream may be applied to introitus for thirty minutes and wiped clean and dried prior to vulvar laser therapy. Patients will be recommended to avoid coital sexual activity for at least 3 days after each laser application because a mild inflammatory reaction may last up to 48 hours after laser therapy. Topical lidocaine 5% ointment may be used for any vulvar pain post-procedure.

Post Treatment Instructions

* Each subject shall be evaluated immediately post-treatment for complications and side effects, excessive bleeding, symptomatic vaginal discharge, pain, etc.
* Each study subject will be asked to assess discomfort of treatment using a 5-point Likert scale.
* The patient will be instructed on the specific activity limitations following the procedure, sedentary activities are recommended for a least a few days.
* The subject will not engage in vigorous exercise or contact sports for at least 72 hours, or until approved by the physician.
* The subject will refrain from douching for at least 72 hours after the procedures.
* Subjects will not engage in intercourse for at least 72 hours post procedure.
* The subject may shower but may not bathe the day following the procedure. They will use regular shower gel or soap.

Vaginal Estrogen Protocol The women in the vaginal estrogen group will be prescribed and asked to administer the conjugated estrogen cream 0.5 g of cream (equivalent to 0.625 mg of conjugated estrogen) intravaginally daily for two weeks (fourteen days) then twice weekly for 24 ± 2 additional weeks.

Vaginal examinations Vaginal Health Index (VHI) score including vaginal pH will be obtained using litmus paper during baseline and each follow-up examination and recorded. This will be obtained during baseline, 6 week, 3 month, and 6 month follow-up by a blinded examiner prior to assessment of vaginal wall elasticity with silastic dilators. A limited vaginal exam will be performed to assess the condition of the vaginal area. This exam will include a vaginal calibration, performed with a standard vaginal dilator (Syracuse Medical). The investigator will determine the largest dilator of the five sizes available (XS, S, M, L, XL), that the subject can comfortably have placed in her vagina. The subject then assesses how much pain she is experiencing when the dilator is placed in her vagina, using a 5-point Likert scale.

* GSM symptom (vaginal dryness, vaginal burning, vaginal itching, dysuria) will be assessed using the VAS.
* Patient evaluation of the overall treatment (PGI) using a 5-point Likert scale will be conducted at 6 week, 3 month and 6 month follow-up visits.
* After each treatment, the PI or co-investigator will be asked to evaluate the ease of treatment using a 5-point Likert scale.
* After each treatment, the subject will be asked the degree of discomfort experienced as a result of treatment using a 5-point Likert scale.
* Events will be evaluated and recorded.

Questionnaires and evaluations Questionnaires will be administered by a research nurse coordinator who is blinded to the patient's therapy. Sexual function, GSM, and urinary function will be evaluated with the 10- cm VAS, Female Sexual Function Index (FSFI), Day-to-day Impact of Vaginal Aging (DIVA), and Urogenital Distress Inventory (UDI-6), both at baseline prior to 1st laser treatment or commencing with vaginal estrogen (depending on treatment group), and at 12 weeks from baseline (+/- 1week) but prior to 3rd laser treatment (if applicable), and at 3 months follow-up after 3rd laser treatment (if applicable). Note that all patients will follow up 6 months from baseline visit for final assessment.

The DIVA questionnaire will be administered at baseline, 3 month, and 6 month follow-up visit period, in addition to the FSFI, UDI-6, VHI, and PGI during final assessment.

Data Collection & Management:

Baseline data will include the following:

* Patient age, race, vaginal parity, menopausal state, BMI, history of previous use of vaginal estrogen
* FSFI, DIVA, and UDI-6 questionnaires
* VAS for GSM symptoms and VHI for objective GSM findings

Data points recorded during the procedure will include:

* Likert Scales for physician assessment of patient comfort during the procedure.
* Adverse events including inability to complete the procedure due to discomfort or constricted vagina

Post-procedure data will include the following:

* The rate of satisfaction of patients with treatment by mean of the Patient Global Impression of Improvement (PGI), using a 5-point Likert scale.
* The degree of difficulty encountered by the physician in performing the treatment, by mean of a 5-point Likert scale.
* Additionally, untoward side effects of treatment such as new bothersome vaginal irritation and significant vaginal bleeding will be recorded.

Protection of each subject's personal health information will be a priority in this study. One master Excel file containing subject personal information including name and medical record number will be kept in a password-protected file, on a designated protected research drive on a password-protected computer in a locked office at each respective institution. In that file, each subject will be assigned a subject identification number that will be used for the purposes of data collection in order to de-identify subjects.

All paper forms used for data collection will be kept in a research cabinet dedicated to this project, which will be locked at all times, in a locked office at the Cleveland Clinic (or other institution name). All forms will contain de-identified information. Identification numbers will correspond to the subjects listed in the master excel file.

All study data will be transferred and managed electronically using REDCap (Research Electronic Data Capture). Each subject will be entered into REDCap using the assigned identification number from the master excel file.

ELIGIBILITY:
Inclusion Criteria:

* Menopausal with absence of menstruation for at least 12 months
* Presence of vaginal atrophy symptoms [subjective assessment of vaginal dryness >7cm on VAS)
* Prolapse stage < II, according to the pelvic organ prolapse quantification (POP-Q) system[31]
* No pelvic surgery within 6 months prior to treatment (vulva biopsy may be included after 2 weeks)
* Understanding and acceptance of the obligation to return for all scheduled follow-up visits

Exclusion Criteria:

* Personal history of vulvovaginal condyloma,,vaginal intraepithelial neoplasia (VAIN), vaginal carcinoma, lichen sclerosis, lichen planus, history of vaginal radiation, history of cervical cancer, other gynecologic cancer, or pelvic radiation
* Acute or recurrent urinary tract infection (UTI), or genital infection (e.g. bacterial; vaginosis, herpes genitalis, candida).
* Personal history of Scleroderma
* Any serious disease, or chronic condition, that could interfere with the study compliance
* Previously undergone reconstructive pelvic surgery within the past 6 months
* Previously undergone reconstructive pelvic surgery with transvaginal mesh kits and sacrocolpopexy with synthetic mesh for prolapse, excluding synthetic slings (unless current untreated exposure or extrusion)
* Have used vaginal estrogen cream, ring or tablet within 1 month prior to entering the study
* Vaginal moisturizers, lubricants or homeopathic preparations within 2 weeks of therapy
* Personal history of thrombophlebitis
* Personal history of heart failure or myocardial infarction within 12 months of procedure
* Use or anticipated use of antiplatelet therapy, anticoagulants, thrombolytics, vitamin E or nonsteroidal anti-inflammatory drugs within 2 weeks pre-treatment
* Taking medications that are photosensitive
* Contraindication to Vaginal Estrogen Therapy
* Unwilling to Take Vaginal Estrogen
* Inability to give informed consent

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2016-03; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marie F Paraiso, M.D., Principal Investigator — The Cleveland Clinic
Locations (6):
- United States (6):
  - Stanford University, Stanford, California
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Christ Hospital, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Brown Medical School, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Ippolito GM, Crescenze IM, Sitto H, Palanjian RR, Raza D, Barboglio Romo P, Wallace SA, Orozco Leal G, Clemens JQ, Dahm P, Gupta P. Vaginal lasers for treating stress urinary incontinence in women. Cochrane Database Syst Rev. 2025 Jul 25;7(7):CD013643. doi: 10.1002/14651858.CD013643.pub2. PMID 40709601
- [Derived] Paraiso MFR, Ferrando CA, Sokol ER, Rardin CR, Matthews CA, Karram MM, Iglesia CB. A randomized clinical trial comparing vaginal laser therapy to vaginal estrogen therapy in women with genitourinary syndrome of menopause: The VeLVET Trial. Menopause. 2020 Jan;27(1):50-56. doi: 10.1097/GME.0000000000001416. PMID 31574047

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CO2 Fractionated Vaginal Laser | Estrogens, Conjugated (USP)
Started | 35 | 34
Completed | 33 | 29
Not Completed | 2 | 5
Not completed — Withdrawal by Subject | 2 | 5

BASELINE CHARACTERISTICS:
Population: Patients were included if they were menopausal with absence of menstruation for at least 12 months with reported presence of vaginal atrophy symptoms (subjective assessment of vaginal dryness greater than or equal to 7cm on visual analog scale (VAS).
Groups:
- Total: Total of all reporting groups
Arm/Group | CO2 Fractionated Vaginal Laser | Estrogens, Conjugated (USP) | Total
Number analyzed (Participants) | 35 | 34 | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (8) | 60 (7) | 61 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 34 | 69
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 32 | 32 | 64
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
BMI [Mean (Standard Deviation); unit: kg/m2] | 25.1 (4.7) | 25.8 (4.4) | 25.4 (4.6)
Parity [Mean (Full Range); unit: pregnancies] | 2 [0 to 6] | 1 [0 to 4] | 2 [0 to 6]
Menopausal [Count of Participants; unit: Participants] | 35 | 34 | 69
Exogenous Hormone Use [Count of Participants; unit: Participants] | 29 | 26 | 55
Vaginal Estrogen Use [Count of Participants; unit: Participants] | 26 | 27 | 53

OUTCOME MEASURES:

1. Primary Outcome: Vaginal Dryness
Description: Vaginal dryness was assessed using a score of 0 (minimum) and 10 (maximum) on a Visual Analog Scale (VAS). Data presented is the mean difference before and after treatment. A higher mean difference signifies that the vaginal dryness score decreased to a greater measure hence resulting in a better outcome.
Time Frame: 6 months
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | CO2 Fractionated Vaginal Laser | Estrogens, Conjugated (USP)
Number analyzed (Participants) | 33 | 29
units on a scale | -5.48 [-8.16 to -2.80] | -5.76 [-8.24 to -3.28]

2. Secondary Outcome: Objective Evaluation of Vaginal Atrophy/Estrogenization
Description: Vaginal health index (VHI) score is measured on a scale of 0 (minimum) to 5 (maximum) and higher scores means a better outcome.
Time Frame: 6 months
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | CO2 Fractionated Vaginal Laser | Estrogens, Conjugated (USP)
Number analyzed (Participants) | 33 | 29
units on a scale | 0.9 [0.2 to 1.6] | 1.2 [0.3 to 2.1]

3. Secondary Outcome: Effect of GMS Symptoms on Quality of Life
Description: DIVA scores are based on a scale of 0 (minimum) to 20 (maximum) with higher scores representing worse outcomes. The data presented are mean differences before and after treatment.
Time Frame: 6 months
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | CO2 Fractionated Vaginal Laser | Estrogens, Conjugated (USP)
Number analyzed (Participants) | 33 | 29
units on a scale | -3.3 [-6.5 to -0.1] | -4.4 [-7.5 to -1.3]

4. Secondary Outcome: Effect of Treatment on Vaginal Maturation Index
Description: Vaginal Maturity Index (VMI) scores are from 0 (minimum) to 100 (maximum) with higher scores representing higher maturity which is a favorable (better) outcome. The results reported are the difference between 2 time points (baseline and 6 month follow up). A change in outcome which is negative signifies a worse outcome. Conversely, a positive change signifies improvement.
Time Frame: 6 months
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | CO2 Fractionated Vaginal Laser | Estrogens, Conjugated (USP)
Number analyzed (Participants) | 33 | 29
units on a scale | 3.9 [-26.7 to 34.5] | 25 [2.4 to 47.6]

5. Secondary Outcome: Vaginal Wall Elasticity Assessed by Number of Participants Able to Tolerate a Larger Vaginal Dilator Size
Description: Participants who were able to tolerate a larger dilator size compared to before treatment (representing improvement in vaginal wall elasticity) were marked as "yes" and participants who could not tolerate a larger size (representing no change in vaginal elasticity) were marked as "no".
Time Frame: 6 months
Population: The data above are represented in tabular form.
Measure: Count of Participants; unit: Participants
Arm/Group | CO2 Fractionated Vaginal Laser | Estrogens, Conjugated (USP)
Number analyzed (Participants) | 33 | 29
Participants | 16 | 17

6. Secondary Outcome: Effect of Treatment on Female Sexual Function
Description: Female Sexual Function Index (FSFI) scores are on a scale of 0 (minimum) to 36 (maximum) with higher scores representing more favorable outcomes. The scores represent the difference between baseline and 6 month follow up. A negative difference signifies worsened function whereas a positive difference signifies improvement.
Time Frame: 6 months
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | CO2 Fractionated Vaginal Laser | Estrogens, Conjugated (USP)
Number analyzed (Participants) | 33 | 29
units on a scale | 1.7 [-5.0 to 8.4] | 4.9 [-3.4 to 13.2]

7. Secondary Outcome: Effect of Treatment on Urinary Symptoms
Description: Urogenital distress inventory (UDI-6) is measures on a scale of 0 (minimum) to 75 (maximum) with higher scores representing less favorable outcomes (more severe urinary symptoms). Data here are presented as mean differences from before and after treatment.
Time Frame: 6 months
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | CO2 Fractionated Vaginal Laser | Estrogens, Conjugated (USP)
Number analyzed (Participants) | 33 | 29
units on a scale | -9.4 [-25.1 to 6.3] | -6.2 [-18.2 to 5.8]

8. Secondary Outcome: Rate of Satisfaction of Patients With Treatment
Description: Patient global impression of improvement (PGI) is a 5-point Likert scale evaluating patient satisfaction after treatment. The 5-point Likert scale for satisfaction indicates 1(Very dissatisfied), 2(Dissatisfied), 3(Same), 4(Satisfied) or 5(Very satisfied). As reported, the responses for level of dissatisfaction after treatment on the Patient Global Index included responses of very dissatisfied and dissatisfied. This is directly out of the questionnaire given to the patient to complete.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | CO2 Fractionated Vaginal Laser | Estrogens, Conjugated (USP)
Number analyzed (Participants) | 33 | 29
Participants
  Better or much better | 24 | 24
  Satisfied or very satisfied | 25 | 22
  Dissatisfied | 3 | 2

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | CO2 Fractionated Vaginal Laser | Estrogens, Conjugated (USP)
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/29
Other Adverse Events (participants affected / at risk) | 5/33 | 5/29
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CO2 Fractionated Vaginal Laser (N=33) | Estrogens, Conjugated (USP) (N=29)
Vaginal bleeding (Reproductive system and breast disorders) | 2 (2) | 2 (2)
Pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Discharge (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Breast Tenderness (Reproductive system and breast disorders) | 0 (0) | 1 (1)
UTI (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 1 (1)
Abdomial cramping (Reproductive system and breast disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-16): https://cdn.clinicaltrials.gov/large-docs/36/NCT02691936/Prot_SAP_000.pdf